CLINICAL TRIAL: NCT04477252
Title: Mobile App as a Guide to Lumbopelvic Stability Exercises in Patients With Chronic Stroke: a Pilot Study of a Randomized Clinical Trial
Brief Title: Mobile App as a Guide to Exercises for Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Neurorehabilitación (Other)
Responsible Party: Principal Investigator, Carina Francisco Salgueiro, Principal Investigator, Clínica de Neurorehabilitación
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIS-2020-02; CORE-app (Other: Clinica de Neurorehabilitación)
Record Dates: First submitted 2020-06-30; First posted 2020-07-20 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Telerehabilitation; Stroke Sequelae; Therapeutic Adherence and Compliance; Mobile Phone Use; Physical Disability; Neurologic Disorder
Keywords: Mobile Applications; Telerehabilitation; Stroke; Therapeutics; Functional recovery; Neurorehabilitation
MeSH Terms: conditions — Treatment Adherence and Compliance; Cell Phone Use; Nervous System Diseases; Stroke

STUDY DESIGN:
Intervention Model Description: In this simple blind randomized controlled pilot study, participants will be recruited from users of the rehabilitation center where the study will be carried out (Neurorehabilitation Clinic - Sant Cugat del Vallés). 30 participants will be recruited. In the recruitment process, patients will be informed about the study, they will be asked to sign an informed consent and the randomization between the experimental group and the control group will be done by computerized program and with the following interventions
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The therapist responsible for the conventional treatment of the patient and the therapist who performs the assessment will not have access to information about the study group the patient encounters. Since the randomization of patients, access to the intervention of the Experimental Group will be facilitated by the researcher on an occasion other than the initial assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App group (Experimental): Use of the Mobile App for the daily performance (Monday to Friday) of lumbopelvic stability exercises apart from the usual physiotherapy treatment for 3 months.
  Interventions: Device: App-core
- conventional physiotherapy (Active Comparator): usual physiotherapy treatment for 3 months
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: App-core — Farmalarm App of the Inmovens group - Vall d´Hebrón Hospital will be used, adapted and updated by the main researcher. The App will have the "rehabilitation" option where the user can consult the description of the exercise and view a demonstration video so that it can be carried out correctly at home, independently or with help. The administrator therapist of the App has the permission to create users, contact them directly through chat or video-call and personalize the exercise program.
  The exercises that will be carried out in this study phase, are described in previous studies by the author Rosa Cabanas et al. All possible exercises will be included in the administration platform, and according to of each user, the prescription of some exercises or others will be made.
  Arms: App group
Other: Conventional physiotherapy — Conventional physiotherapy is considered neuromotor development therapy as the most frequently used therapy in the management of stroke patients and in the center where the study is performed.
  Arms: conventional physiotherapy

SUMMARY:
Introduction: Stroke continues to be one of the leading causes of disability in the Spanish adult population with the presentation of impairments such as alteration of mobility and a consequent reduction in quality of life. These sequelae, generally chronic, generates a significant expense and saturation of social and health services. With the growth in the number of cases, the development of new rehabilitation approaches and updating of the social context becomes pertinent, such as the incorporation of telerehabilitation to assist individuals with stroke.

Objectives: To analyze adherence to physical rehabilitation by mobile App and to evaluate the effectiveness of lumbopelvic stability exercises performed at home with the App.

Material and methods: Randomized controlled single blind pilot study (n = 30). Participants with Stroke (<6 months) will be randomized between two groups (App for carrying out lumbopelvic stability exercises + usual treatment versus usual treatment). The study will last 3 months and App adherence, Quality Of Life, participation in Daily Life, functionality, sitting balance, standing balance and gait will be taken as variables.

Expected results: It is thought that the use of an App can contribute to rehabilitation in its chronic phase, monitorization and fallow-up the clinical evolution of the patient. Even if chronicity leads us to think about the stabilization of the physical condition, It is thought that the best results will be found among the subjects who will use the App.

DETAILED DESCRIPTION:
The recruitment of participants will be done in a personalized way through a verbal invitation from the responsible therapist.

The therapists of the center will be informed about the inclusion criteria in this study in order to proceed with the personalized invitation.

In the case that the participant meet the inclusion criteria and wishes to participate in the study, the professional evaluator is contacted to begin the process of submission in this study.

The professional evaluator has the responsibility to explain to the participant what the study consists of The professional evaluator is responsible for giving the participant the study information sheet (approved by the ethics committee and the management of the center where the study will be conducted).

The professional evaluator is responsible for collecting the signature of the informed consent to participate in this study (approved by the ethics committee and the management of the center where the study will be conducted).

A numerical code (from 1 to 30) will be assigned to each patient according to the order of recruitment to keep their identity secret.

The code attributed to each participant will appear in the individual data collection notebook The association between the participant's identity and the attributed code will be known by the professional evaluator The code attributed to each participant will be entered in the spreadsheet where the collected data and results of the assessment tests will be uploaded.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of stroke with cortical or subcortical, ischemic or hemorrhagic involvement with more than 6 months of evolution
* Clinical symptoms of hemiplegia or hemiparesis
* Over 18 years of age
* Ability to understand and execute simple instructions
* Score equal to or less than 10 in the Spanish version of the Trunk Impairment Scale 2.0
* Be a frequent user of smartphone or tablet. Failing this, the direct family member / caregiver is considered.

Exclusion Criteria:

* Appearance of any disease or aggravation of any of the comorbidities that the patient presents that prevents rehabilitation (example: dialysis)
* Suffer a second episode of Stroke.
* Fractures in any of the lower extremities or important structural alterations in the trunk.
* Death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence: Scale of System Uses | week 12
  Adherence to the use of the mobile App using Scale of System Uses. Minimum Score:0 Maximum Score: 100 (higher scores mean a better result)
Adherence: Administration panel of the App | week 12
  Adherence to the use of the mobile App using the data extracted by the administration panel of the App. Consider 5 days / week the optimal use (100%) and a total use of 0 to 20 days in 12 weeks will be considered low adherence (0-33%), 21 to 41 days (33-66%) regular adherence and 42 to 60 days (66-100% :) good adherence.

OTHER OUTCOMES:
Quality of Life: EuroQol test | 0, 6, 12 weeks
  Quality of Life using EuroQol 5d5l. This questionnaire is made up of two parts. Part I: One part with 5 questions scored from 1 to 5 (1 represents absence of problem and 5 the absolute limitation). The total score ranges from 5 to 25 in which higher results represent a worse outcome.
  Part II: Consisting of a numerical scale from 0 to 100 on the general state of health, in which 0 represents the worst level of health and 100 the best level of health that individuals can perceive.
Participation in Activity of Daily Living: Barthel Index | 0, 6, 12 weeks
  Participation in Activity of Daily Living using Barthel Index Scale. Minimum Score: 0; Maximum Score: 100. Higher score means better outcomes
Functionality: Rankin scale | 0, 6, 12 weeks
  Functionality using Rankin Scale. Minimum Score: 0; Maximum Score: 6. Higher score means worse outcomes
Sitting balance: Spanish versions of the Trunk Impairment Scale 2.0 | 0, 6, 12 weeks
  Sitting balance using Spanish versions of the Trunk Impairment Scale 2.0. Minimum Score: 0; Maximum Score: 26. Higher score means better outcomes
Sitting balance: Function in Sitting Test | 0, 6, 12 weeks
  Sitting balance using Function in Sitting Test. Minimum Score: 0; Maximum Score: 56. Higher score means better outcomes
Standing balance: Berg Balance Scale | 0, 6, 12 weeks
  Standing balance using Berg Balance Scale. Minimum Score: 0; Maximum Score: 56. Higher score means better outcomes
Standing balance: Spanish version of the Postural Assessment Scale for stroke patients | 0, 6, 12 weeks
  Standing balance using Spanish version of the Postural Assessment Scale for Stroke patients. Minimum Score: 0; Maximum Score: 36. Higher score means better outcomes
G-Walk accelerometer system: Duration of double and individual support | 0, 6, 12 weeks
  Duration of double and individual support (%). The software provides the values from subjects and the mean values of the population. It will be take into account the difference between the subject values and the mean in the population without pathology. Higher scores means worse results.
G-Walk accelerometer system: Duration of support and swing gait phases from right anda left lower limb | 0, 6, 12 weeks
  Duration of support and swing gait phases from right anda left lower limb(%). The software provides the values from subjects and the mean values of the population. It will be take into account the difference between the subject values and the mean in the population without pathology. Higher scores means worse results.
G-Walk accelerometer system: Cadence of stride | 0, 6, 12 weeks
  Cadence of stride (steps/minutes). The software provides the values from subjects and the mean values of the population. It will be take into account the difference between the subject values and the mean in the population without pathology. Higher scores means worse results.
G-Walk accelerometer system: Gait speed | 0, 6, 12 weeks
  Gait speed (metres/second).The software provides the values from subjects and the mean values of the population. It will be take into account the difference between the subject values and the mean in the population without pathology. Higher scores means worse results.
G-Walk accelerometer system: Step length | 0, 6, 12 weeks
  Step length (%). The software provides the values from subjects and the mean values of the population. It will be take into account the difference between the subject values and the mean in the population without pathology. Higher scores means worse results.
G-Walk accelerometer system | 0, 6, 12 weeks
  Stride length (meters). The software provides the values from subjects and the mean values of the population. It will be take into account the difference between the subject values and the mean in the population without pathology. Higher scores means worse results.
number of falls in the last six weeks | 0, 6, 12 weeks
  Balance. Higher scores means worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Carina F Salgueiro, MSc, Principal Investigator — Clínica de Neurorehabilitación
Locations (1):
- Clinica de neurorehabilitacion SL, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
It is intended to share the data with other researchers such as the statistical team through encrypted e-mail.

REFERENCES:
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Brewer L, Horgan F, Hickey A, Williams D. Stroke rehabilitation: recent advances and future therapies. QJM. 2013 Jan;106(1):11-25. doi: 10.1093/qjmed/hcs174. Epub 2012 Sep 27. PMID 23019591
- [Background] Schmid AA, Van Puymbroeck M, Altenburger PA, Miller KK, Combs SA, Page SJ. Balance is associated with quality of life in chronic stroke. Top Stroke Rehabil. 2013 Jul-Aug;20(4):340-6. doi: 10.1310/tsr2004-340. PMID 23893833
- [Background] Isho T, Usuda S. Association of trunk control with mobility performance and accelerometry-based gait characteristics in hemiparetic patients with subacute stroke. Gait Posture. 2016 Feb;44:89-93. doi: 10.1016/j.gaitpost.2015.11.011. Epub 2015 Nov 26. PMID 27004638
- [Background] Cabanas-Valdes R, Bagur-Calafat C, Girabent-Farres M, Caballero-Gomez FM, Hernandez-Valino M, Urrutia Cuchi G. The effect of additional core stability exercises on improving dynamic sitting balance and trunk control for subacute stroke patients: a randomized controlled trial. Clin Rehabil. 2016 Oct;30(10):1024-1033. doi: 10.1177/0269215515609414. Epub 2015 Oct 8. PMID 26451007
- [Background] Cabanas-Valdes R, Bagur-Calafat C, Girabent-Farres M, Caballero-Gomez FM, du Port de Pontcharra-Serra H, German-Romero A, Urrutia G. Long-term follow-up of a randomized controlled trial on additional core stability exercises training for improving dynamic sitting balance and trunk control in stroke patients. Clin Rehabil. 2017 Nov;31(11):1492-1499. doi: 10.1177/0269215517701804. Epub 2017 Mar 29. PMID 28351168
- [Background] Cabanas-Valdes R, Cuchi GU, Bagur-Calafat C. Trunk training exercises approaches for improving trunk performance and functional sitting balance in patients with stroke: a systematic review. NeuroRehabilitation. 2013;33(4):575-92. doi: 10.3233/NRE-130996. PMID 24018373
- [Background] Chen Y, Abel KT, Janecek JT, Chen Y, Zheng K, Cramer SC. Home-based technologies for stroke rehabilitation: A systematic review. Int J Med Inform. 2019 Mar;123:11-22. doi: 10.1016/j.ijmedinf.2018.12.001. Epub 2018 Dec 11. PMID 30654899
- [Background] Zhou X, Du M, Zhou L. Use of mobile applications in post-stroke rehabilitation: a systematic review. Top Stroke Rehabil. 2018 Sep 13:1-11. doi: 10.1080/10749357.2018.1482446. Online ahead of print. PMID 30209991
- [Background] Sanchez Rodriguez MT, Collado Vazquez S, Martin Casas P, Cano de la Cuerda R. Neurorehabilitation and apps: A systematic review of mobile applications. Neurologia (Engl Ed). 2018 Jun;33(5):313-326. doi: 10.1016/j.nrl.2015.10.005. Epub 2015 Dec 17. English, Spanish. PMID 26703120

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT04477252/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT04477252/ICF_000.pdf